CLINICAL TRIAL: NCT04877015
Title: Vibrotactile Coordinated Reset: A Non-invasive Treatment for Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stanford terminated the study with no reason given.
Sponsor: Synergic Medical Technologies, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 59621
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Vibrotactile Coordinated Reset (vCR) (Active Comparator): Participants in this arm will receive active vCR stimulation.
  Interventions: Device: Active Vibrotactile Coordinated Reset (vCR)
- Sham Vibrotactile Coordinated Reset (vCR) (Sham Comparator): Participants in this arm will receive sham vCR stimulation.
  Interventions: Device: Sham Vibrotactile Coordinated Reset (vCR)

INTERVENTIONS:
Device: Active Vibrotactile Coordinated Reset (vCR) — Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. A specific pattern of vibration to each fingertip is delivered which theoretically disrupts abnormal synchrony in the brain.
  Other Names: VT Brain Glove
  Arms: Active Vibrotactile Coordinated Reset (vCR)
Device: Sham Vibrotactile Coordinated Reset (vCR) — Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. An inactive pattern of vibration to each fingertip is delivered which theoretically will not have the effects of active vCR.
  Other Names: VT Brain Glove
  Arms: Sham Vibrotactile Coordinated Reset (vCR)

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on motor ability within Parkinson's patients. vCR will be administered with a device called the VT Brain Glove. vCR is expected to provide patients with a non-invasive alternative to the most widely used treatments such as levodopa and or deep brain stimulation. This study will include a dedicated sham that will aid in understanding true treatment effects from vCR.

DETAILED DESCRIPTION:
Current treatments for Parkinson's disease include medications, surgical measures, or a combination of both. However, long term use of medications can result intolerable side effects, especially at higher doses. If patients under go Deep Brain Stimulation (DBS) surgery, risks include risk of stroke, infection, seizure, hemorrhage or others we may not anticipate. Our investigators hope to confirm a non-invasive method of applying the stimulation by vibrotactile stimulation delivered through the fingertips will alleviate severity in motor symptoms in Parkinson's patients

ELIGIBILITY:
1. Between the ages of 45-85
2. Diagnosis of idiopathic Parkinson's disease
3. Bilateral impairment, as defined as Hoehn & Yahr Stages II-IV in the on-medication state
4. Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III motor improvement greater than or equal to 30% when on medication compared to when off medication.
5. Participants must be on stable dose of dopaminergic medication for 1 month prior to baseline visit.
6. Able to provide informed consent.
7. Appropriate social support if required during an off state.
8. Comfortable with technology; can use a computer, check email, and access the internet; can initiate and engage in a virtual meeting for training and monitoring purposes.
9. Participants must speak English and can communicate with staff without the need of an interpreter.
10. If patient is on medication that affects brain function or alters EEG activity, the patient must feel comfortable going off this medication prior to EEG recordings

Exclusion Criteria

1. Presence of other forms of non-idiopathic parkinsonism, including but not limited to atypical parkinsonism, medication-induced parkinsonism, and vascular parkinsonism.
2. Presence of other brain diseases (i.e. major depression, dementia, Attention Deficit/Hyperactivity Disorder (ADHD) psychosis, etc…).
3. Severe depression, severe anxiety, or severe psychosis for the purpose of excluding candidates at an elevated risk of suicidal tendencies.
4. Participation in another drug, device, biologic, or intervention trial concurrently or within the preceding 30 days.
5. Physical limitations unrelated to Parkinson's disease.
6. Speech problems or excessive drooling so severe patient cannot communicate properly to staff.
7. Presences of dopamine dysregulation syndrome.
8. On dopamine agonist(s) and exhibits compulsive behaviors.
9. Current delirium
10. Pregnancy, breastfeeding, or trying to get pregnant during the duration of the study.
11. History of epilepsy or traumatic brain injury.
12. Brain surgery (i.e. DBS implantation) or craniotomy.
13. Neurostimulator.
14. A type of hairstyle that would impede the use of a EEG cap
15. Severe sensory abnormalities of the fingertips such as vibratory urticaria.
16. Current or ongoing hallucinations, delusions.
17. The PI and study's neurologist deems the patient ineligible.
18. Patient has a functional movement disorder that prevents accurate Parkinson's disease evaluations

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 | 14months
  This scale measures motor ability within Parkinson's patients. For part 3, the scales minimum values is 0 and max value is 132. Higher scores indicate more impaired motor ability, while lower scores indicate less impaired motor ability. A score of 0 indicates no motor impairment. This evaluation will be done in person at baseline, 3,6 and 7 months. The remote version will be done at 10, 13 and 14 months

SECONDARY OUTCOMES:
Spontaneous electroencephalography (EEG) | 7 months
  Spontaneous EEG is recorded at baseline, 3, 6 and 7 months. 3 types of recordings will occur per visit:5 minute Baseline, 16 minute during vibrotactile therapy (sham or active vCR depending on the participant group) and post vibrotactile therapy. Power spectral density (PSD) will be calculated from source constructed EEG activity for each frequency band of interest (Delta: 2-4 Hz; Theta: 5-7 Hz; Alpha: 8-12 Hz; Low Beta: 13-16 Hz; Mid Beta: 17-20 Hz; High Beta: 21-30 Hz; and Gamma: 31-50 Hz) using the Welch method with a 2-s window overlapping by 50%. Relative power (RP) is calculated by taking the sum of each frequency band and dividing it by the total power across the spectrum (2-50 Hz).
Sensorimotor task EEG | 7 months
  Sensorimotor activity during the EEG will be recorded at baseline, 3, 6 and 7 months. Patients receive a single vibratory stimulus to a random finger (excluding the thumb) on their left or right hand and are instructed with their non-stimulated hand to push the response button as fast as possible when they feel the vibratory burst. Each finger receives an equal number of vibratory pulses (50 per finger, equaling 200 trials per hand) in a randomized order. Cortically, we expect to look at motor evoked potentials in response to cued vibration by means of their amplitude (micro-volts) and latency (time in milliseconds) and their changes throughout the course of treatment. Reaction time (in milliseconds) will also be documented.
Vibration-only evoked EEG potentials | 7 months
  We will record vibration-only evoked EEG potentials at baseline, 3, 6 and 7 months.We will look at how single vibratory pulses to each finger (excluding the thumb) affect different motor and sensory areas of the brain.Each finger receives an equal number of vibratory pulses (50 per finger, equaling 200 trials per hand) in a randomized order. Cortically, we expect to look at sensory evoked potentials in response to vibration by means of their amplitude (micro-volts) and latency (time in milliseconds) and their changes throughout the course of treatment.
PD Quality of Life Questionnaire-39 (PDQ-39) | 14 months
  The PD Quality of Life Questionnaire-39 (PDQ-39) is a self-report questionnaire that examines health related difficulties specific to PD in eight quality of life categories within the last month. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100, with higher % indicating more health problems. This questionnaire will be taken at baseline, 3, 6, 7, 10, 13 and 14 months.
Parkinson's disease sleep scale (PDSS) | 14 months
  The Parkinson's disease sleep scale (PDSS) is a visual analogue scale addressing 15 commonly reported symptoms associated with sleep disturbance in the past week. The scores for each item range from 0 (symptom severe and always experienced) to 10 (symptom-free). The maximum cumulative score for the PDSS is 150 This questionnaire will be taken at baseline, 3, 6, 7, 10, 13 and 14 months.
University of Pennsylvania Smell Identification Test (UPSIT) | 7 months
  University of Pennsylvania Smell Identification Test (UPSIT) is a smell test comprised of 40 odors, in which patients try to correctly identify the odor presented. The test is a forced choice paradigm, that is, if an individual is unsure of an answer they are forced to guess a response hence a score of 25% on average would reflect random guessing. An UPSIT result is scored out of 40 where a higher score indicates better olfaction.This test will be taken at baseline, 3, 6, and 7 months
Vibratory temporal discrimination task (VTDT) | 7 months
  The vibratory temporal discrimination task (VTDT) consists of two vibratory bursts, with one burst delivered to the index finger and one burst to the middle finger. This procedure will be performed on the right and left hand separately. The patient is instructed to judge if he/she felt a delay between the two vibratory bursts. This task was designed as a possible calibration method for future vCR studies by serving as a sensitivity measure for vibratory temporal changes, in which reduced perceived vibratory time differences (in milliseconds) correspond to increased vibratory temporal discrimination. This task will be done at at baseline, 3, 6 and 7 months.
Speech and voice assessments | 7 months
  To collect samples, a head-worn, unidirectional microphone will be placed over the participant's ears and the microphone will be adjusted so that it is 6 cm from the participant's mouth. Specific samples will include sustained vowel phonations, sentence and paragraph length reading passages, and spontaneous speech. From these samples, speech and voice assessments will be conducted including measures of articulatory precision, speech intelligibility, speech rate, auditory-perceptual ratings of voice, and acoustic measures of vocal fundamental frequency, vocal intensity, and fundamental frequency and intensity variability. The speech and voice evaluation will be done at baseline, 3, 6 and 7 months
Kinesia One motor evaluation | 14 months
  The Kinesia One motor evaluation, which uses a wearable accelerometer to assess Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3. Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities). Patients will perform this test at baseline, 3, 6,7 months in person and at home at 10, 13 and 14 months.
Levodopa equivalent daily dose (LEDD) | 14 months
  Levodopa equivalent daily dose (LEDD) will measured at baseline, 3,6,7,10,13 and 14 months. LEDD is calculated as a sum of each Parkinson's medication.
Freezing of Gait Questionnaire | 14 months
  The Freezing of Gait Questionnaire (FOGQ) assesses Freezing of Gait (FOG) severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning). The FOG is comprised of 6 questions measured on a 0 to 4 scale (where 0 is normal and 4 represents severe abnormalities). The scores are summed together with 0 representing the best possible score and 24 representing the worst possible score. FOG will measured at baseline, 3,6,7,10,13 and 14 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tass, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Potentially available upon request.

REFERENCES:
- [Derived] Pfeifer KJ, Cook AJ, Yankulova JK, Mortimer BJP, Erickson-DiRenzo E, Dhall R, Montaser-Kouhsari L, Tass PA. Clinical Efficacy and Dosing of Vibrotactile Coordinated Reset Stimulation in Motor and Non-motor Symptoms of Parkinson's Disease: A Study Protocol. Front Neurol. 2021 Nov 18;12:758481. doi: 10.3389/fneur.2021.758481. eCollection 2021. PMID 34867742